CLINICAL TRIAL: NCT05147402
Title: A Phase 1, Single Center, Open Label, Randomized Sequence, 2-period Cross-over Study to Determine the Effect of Food on the Relative Bioavailability of 3,4-methylenedioxymethamphetamine (MDMA) Oral Formulation in Healthy Volunteers
Brief Title: Food Effects on Bioavailability of MDMA in Healthy Volunteers
Acronym: MPKF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPKF
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pharmacokinetics
Keywords: MDMA; Metabolism; Methylenedioxymethamphetamine; midomafetamine
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Participants who are enrolled in the study will be randomized to 1 of 2 dosing regimens, both of which receive the same intervention in opposite order. Group 1 receives a Fasted Treatment followed by a Fed Treatment, while Group 2 receives a Fed Treatment followed by a Fasted Treatment.
Masking Description: No masking; open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasted Treatments with 120 mg midomafetamine HCl (Active Comparator): Following an overnight fast of at least 10 hours, participants will be administered 100 mg midomafetamine (equivalent to 120 mg midomafetamine HCl) with 240 mL of water. No food should be allowed for at least 4 hours post-dose.
  Interventions: Drug: midomafetamine
- Fed Treatments with 120 mg midomafetamine HCl (Active Comparator): A high-fat (approximately 50 percent of total caloric content of the meal) and high-calorie (approximately 800 to 1000 calories) meal will be used as a test meal for food-effect evaluation. Following an overnight fast of at least 10 hours, participants will start the recommended meal 30 minutes prior to administration of the drug product. Participants will eat this entire meal in 30 minutes or less. 100 mg midomafetamine (equivalent to 120 mg midomafetamine HCl) will be administered 30 minutes after start of the meal with 240 mL of water.
  Interventions: Drug: midomafetamine

INTERVENTIONS:
Drug: midomafetamine — 100 mg midomafetamine (equivalent to 120 mg midomafetamine HCl).
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine HCl; MDMA

SUMMARY:
The goal of this clinical trial is to learn if food impacts absorption of MDMA in participants who are either fed or fasted.

The main question it aims to answer is: What is the effect of eating food on the safety of taking oral MDMA?

Researchers will compare participants who are fasted for 10 hours to participants who are fed a high-fat and high-calorie meal.

Participants will be randomized to either the fed or fasted group, then be administered MDMA. Vitals and blood samples will be taken. Then, participants will be assigned to the opposite condition and vitals and blood samples will be taken.

DETAILED DESCRIPTION:
This phase I, open-label, randomized sequence, multi-dose, 2-period crossover pharmacokinetic (PK) study assesses the effect of food on the relative bioavailability of MDMA. In addition, an increase in heart rate is anticipated following MDMA administration. Therefore, the secondary purpose of this study is to evaluate the effect of food on the safety and tolerability of oral MDMA, as well as MDMA effects on ECG.

Potential participants will be identified by the clinical site and invited to phone screen for the study. Following informed consent, potential study participants will undergo screening examinations to assess eligibility for inclusion in the study.

Participants will be randomized to receive one of two conditions before the other:

* Fasted Treatments: 10 hours of fasting followed by MDMA administration with 240 mL water.
* Fed Treatments: A high-fat (approximately 50 percent of total caloric content of the meal) and high-calorie (approximately 800 to 1000 calories) meal will be consumed within 30 minutes of MDMA administration.

Participants will be confined at the Clinical Research Unit (CRU) for each Dosing Session from the time of check-in on the night before dosing until discharge 48 hours after dosing. MDMA will be administered on Day 1 following the treatment sequence to which the participant has been randomized. Concentration-time profiles of MDMA will be determined in the time interval 0-72 hours post-dose, according to the expected PK profiles of MDMA and its metabolites. Participants will remain at the CRU for at least 36 hours after administration of study drug for collection of serial blood samples for PK analysis and safety monitoring. An additional outpatient visit will occur 72 hours after dosing to collect a final PK sample and perform safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Are fluent in speaking and reading the predominantly used or recognized language of the study site.
* Are able to swallow pills.
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 7 days after the last Experimental Session.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have uncontrolled hypertension.
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] corrected by Bazett's formula).
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have evidence or history of significant medical disorders.
* Have symptomatic liver disease.
* Have history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control.
* Are abusing illegal drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve from dosing time to last measurement - Plasma concentration of MDMA | 0 to 1 day after drug administration
  Computed exposure to MDMA using blood collected periodically at pre-dose as well as 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, and 12 hours post drug administration.
Area under the curve from dosing time to last measurement - Plasma concentration of active metabolite MDA | 0 to 1 day after drug administration
  Computed exposure to MDMA using blood collected periodically at pre-dose as well as 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, and 12 hours post drug administration

CONTACTS AND LOCATIONS:
Overall Officials: William B Smith, M.D., Principal Investigator — Alliance for Multispecialty Research
Locations (1):
- Alliance for Multispecialty Research LLC, Knoxville, Tennessee, United States